CLINICAL TRIAL: NCT01416870
Title: Bioequivalence Study of ICI176,334-1 (Bicalutamide New Formulation) in Japanese Healthy Male Subjects - Evaluation of Bioequivalence of ICI176,334-1 and Casodex Tablet (80mg)
Brief Title: Bioequivalence of Bicalutamide New Formulation in Japan
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6874L00012
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Bioequivalence; pharmacokinetics; safety; bicalutamide; Casodex; Japanese; healthy subject
MeSH Terms: interventions — bicalutamide; Tablets

ARMS (3):
- Active 1 (Experimental): 34 subjects will receive ICI176,334-1without water
  Interventions: Drug: ICI176,334-1
- Active 2 (Experimental): 34 subjects will receive ICI176,334-1 with water
  Interventions: Drug: ICI176,334-1
- Active 3 (Experimental): 34 subjects will receive Casodex 80 mg tablet
  Interventions: Drug: Casodex 80 mg tablet

INTERVENTIONS:
Drug: ICI176,334-1 — Subject will receive single dose of ICI176,334-1
  Arms: Active 1; Active 2
Drug: Casodex 80 mg tablet — Subject will receive single dose of Casodex 80 mg tablet
  Arms: Active 3

SUMMARY:
The purpose of this study is to investigate the bioequivalence of Bicalutamide new formation with Casodex commercial tablet (80mg) in Japanese healthy male subjects

DETAILED DESCRIPTION:
Bioequivalence study of ICI176,334-1 (Bicalutamide new formulation) in Japanese healthy male subjects - evaluation of bioequivalence of ICI176,334-1 and Casodex tablet (80mg)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Japanese healthy male subjects aged 20 to 45 years
* Male subjects should be willing to use barrier contraception ie, condoms, until 3 months after the last dose of investigational product
* Have a body mass index (BMI) between 17 and 27 kg/m2
* Eligible based on the physical findings, supine BP, pulse rate, ECG and laboratory assessments, as judged by the investigator(s)

Exclusion Criteria:

* Presence of any disease under medical treatment
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunological, blood, endocrine, neurological or mental disease to interfere with absorption, distribution, metabolism or excretion of drugs judged by investigator(s)
* Presence of any infectious disease, such as bacteria, virus and fungus
* Presence of allergic disorder, such as asthma, pollen disease or atopic dermatitis, and judged as necessary any medical treatment
* Any large surgical history of gastrointestinal tract such as gastric/intestinal resection or suturation

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To investigate the bioequivalence of ICI176,334-1 by assessment of Cmax (Maximum Concentration of drug). | Blood samples are taken repeatedly for 72 hours and also taken occasionally up to 672 hours after each dose period
To investigate the bioequivalence of ICI176,334-1 by assessment of AUC (concentration Area Under the Curve). | Blood samples are taken repeatedly for 72 hours and also taken occasionally up to 672 hours after each dose period
To investigate the bioequivalence of ICI176,334-1 by assessment of t1/2 (half time) of bicalutamide | Blood samples are taken repeatedly for 72 hours and also taken occasionally up to 672 hours after each dose period

SECONDARY OUTCOMES:
To assess the safety by assessment of adverse event. | Subjects will be monitored for adverse events prior to treatment and up to 42 -49 days (follow-up) after the last dose.
To assess the safety by assessment of vital signs. | Subjects will be monitored for vital signs prior to treatment and up to 42 -49 days (follow-up) after the last dose.
To assess the safety by assessment of electrocardiograms (ECGs) | Subjects will be monitored for electrocardiograms(ECGs) prior to treatment and up to 42 -49 days (follow-up) after the last dose.